CLINICAL TRIAL: NCT05729126
Title: The Discrepancy in Radiologists' Practice of Intravenous Contrast Imaging Studies Among Chronic Kidney Disease Patients
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mahmoud Hamada imam, Assisstant professor, Benha University
Other Study IDs: BN-120420
Record Dates: First submitted 2022-08-19; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Chronic Kidney Diseases; Chronic Kidney Disease 5D
Keywords: Chronic kidney disease; Hemodialysis; Intrevenous Contrast
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- active arm: participants responding to the questionnaire emailed.
  Interventions: Other: Questionnare

INTERVENTIONS:
Other: Questionnare — A questionnaire form is emailed to radiologists to get their response of their practice with hemodialysis and chronic kidney disease patients

SUMMARY:
* There is a discrepancy between protocols used for intravenous imaging for chronic kidney disease including hemodialysis patients among different hospitals and even, among radiologists same selves.
* This questionnaire based study aims to quantify that discrepancy and describe the variables associated with the discrepancy.

DETAILED DESCRIPTION:
* There is a discrepancy between protocols used for intravenous imaging for chronic kidney disease including hemodialysis patients among different hospitals and even, among radiologists same selves.
* This questionnaire-based study aims to quantify that discrepancy and describe the variables associated with the discrepancy.

ELIGIBILITY:
Inclusion Criteria:

* Practicing radiologist

Exclusion Criteria:

* retired radiologist

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Radiology physicians
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
time from IV contrast study and next dialysis session | 1 day
  time from IV contrast study and next dialysis session

CONTACTS AND LOCATIONS:
Locations (1):
- Benha Faculty of Medicine, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
For privacy reasons of participants